CLINICAL TRIAL: NCT07165223
Title: A Phase IIIb Clinical Study to Assess the Efficacy and Safety of GZR4 in Subjects With Type 2 Diabetes Mellitus Treated With Basal Insulin
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR4-T2D-304
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Diabetes
Keywords: GZR4 insulin
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR4 group (Experimental)
  Interventions: Drug: GZR4
- insulin Icodec group (Active Comparator)
  Interventions: Drug: Insulin Icodec group

INTERVENTIONS:
Drug: GZR4 — GZR4 s.c., once-weekly，treat-to-target dose
  Arms: GZR4 group
Drug: Insulin Icodec group — insulin Icodec s.c., once-weekly，treat-to-target dose
  Arms: insulin Icodec group

SUMMARY:
This study will be conducted to compare the efficacy, safety and patient-reported outcome of GZR4 and Insulin Icodec with or without Non-Insulin Antidiabetic Agents in subjects with Type 2 Diabetes Mellitus (T2DM) treated with basal insulin.

ELIGIBILITY:
Inclusion Criteria:

* Sign the Informed Consent Form (ICF) before the study, fully understand the contents, process and possible adverse reactions of the study, and be able to follow the contraindications and restrictions specified in this protocol.
* Males and females age ≥ 18 years at the time of informed consent.
* The pregnancy test for β-human chorionic gonadotropin (hCG) must be negative for women of childbearing potential during the screening period and prior to randomization.
* From signing the Informed Consent Form until 3 weeks after the end of treatment, female subjects of childbearing potential and male subjects and their partners must agree to use reliable contraceptive measures and not donate eggs (ova, oocytes) or sperm for assisted reproductive purposes.
* According to the diagnostic criteria and classification of diabetes mellitus issued by the World Health Organization (WHO) in 1999, and the supplementary diagnostic criteria recommended by WHO for diagnosis with Hemoglobin A1c (HbA1c) (2011), the time to diagnose T2DM is ≥ 180 days at screening.
* Before screening, basal insulin was given once or twice a day. Or Insulin Icodec was given once-weeekly before screening.

Exclusion Criteria:

* A history of allergy to drugs with two or more mechanisms of action in the past, or known allergies, hypersensitivity, or intolerance to the investigational medicinal product or its excipients.
* Subjects who are pregnant, lactating or planning to become pregnant during the study at screening.
* Participated in any drug clinical study (received non-placebo medication during the study) within a recent period of time (90 days or 5 half-lives of the previous investigational medicinal product, whichever is longer), or plans to participate in another clinical study before completing all scheduled assessments in this clinical study.
* Underwent invasive cardiovascular or cerebrovascular procedures within 180 days before screening; or experienced acute heart failure, myocardial infarction, stroke, or hospitalization due to angina unstable, transient ischaemic attack, or other acute cardiovascular events within 180 days before screening; or have a history of chronic cardiac failure classified as New York Heart Association Class III or IV at screening; or plan to undergo coronary, carotid, or peripheral arterial revascularisation procedures during the study; or have clinically significant abnormalities on the electrocardiogram (ECG) that the investigator considers inappropriate to participate in this study (such as second-degree type II or third-degree atrioventricular block, ventricular fibrillation, etc.).
* History of malignant tumors within 5 years before screening (excluding adequately treated or resected non-metastatic basal or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer in situ) or the presence of underlying malignancy at screening.
* The patient with SBP ≥ 160 mmHg or DBP ≥ 100 mmHg during screening.
* Subjects who are unable to comply with the requirements of this protocol as judged by the investigator, or have any other conditions that the investigator considers inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to week 26

SECONDARY OUTCOMES:
hypoglycaemia events | From baseline (week 0) to week 26
adverse events | From baseline (week 0) to week 26
Change in weight | From baseline (week 0) to week 26

CONTACTS AND LOCATIONS:
Locations (1):
- Gan & Lee Pharmaceuticals Shandong Co., Ltd., Linyi, Shandong, China